CLINICAL TRIAL: NCT01626170
Title: Observational - Identifying and Validating Novel Mechanisms of Radiation Resistance in Rhabdomyosarcoma
Brief Title: Studying Mechanisms of Radiation Therapy Resistance in Samples From Younger Patients With Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST12B6; NCI-2012-01979 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Alveolar Childhood Rhabdomyosarcoma; Embryonal Childhood Rhabdomyosarcoma; Previously Treated Childhood Rhabdomyosarcoma; Previously Untreated Childhood Rhabdomyosarcoma; Recurrent Childhood Rhabdomyosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative (laboratory biomarker analysis): Archived tissue samples of matched primary-relapsed and non-matched primary are analyzed for genomic DNA, DNA methylation profiles, RNA sequencing, differences between alveolar rhabdomyosarcoma (ARMS) and embryonal rhabdomyosarcoma (ERMS), gene expression profiles, target-of-rapamycin complex 1 (TORC1) and TORC2 pathway intermediates, and paired box 3 (PAX3)/forkhead box O1 (FOXO1) translocation by microarray, immunohistochemical staining, and fluorescence in situ hybridization (FISH).
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This laboratory study is looking into mechanisms of radiation therapy resistance in samples from younger patients with rhabdomyosarcoma. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer

DETAILED DESCRIPTION:
Observational Study Model: Cohort Time Perspective: Retrospective Biospecimen Retention: Samples with DNA Biospecimen Description: Tissue Study Population Description: Primary care clinic Sampling Method: Non-probability sample

OBJECTIVES:

I. Determine the molecular response/resistance signatures with radiotherapy and standard chemoradiation treatments using the xenograft model of the Pediatric Preclinical Testing Program (PPTP).

II. Validate these novel pathways/biomarkers by their detection within clinically annotated patient tumor tissue samples and testing their associations with clinical response, local control rates, and overall survival rates.

OUTLINE: Archived tissue samples of matched primary-relapsed and non-matched primary are analyzed for genomic DNA, DNA methylation profiles, RNA sequencing, differences between alveolar rhabdomyosarcoma (ARMS) and embryonal rhabdomyosarcoma (ERMS), gene expression profiles, target-of-rapamycin complex 1 (TORC1) and TORC2 pathway intermediates, and paired box 3 (PAX3)/forkhead box O1 (FOXO1) translocation by microarray, immunohistochemical staining, and fluorescence in situ hybridization (FISH).

ELIGIBILITY:
Inclusion Criteria:

* Tissues requested from the Children Oncology Group (COG) sarcoma banking protocol COG-D9902
* All subtypes of rhabdomyosarcoma specimens

  * Matched primary-relapsed specimens (from same patient, separated by time):

    * Frozen tissue if available
    * Scrolls of formalin-fixed paraffin-embedded tissue (if frozen not available)
    * 10 unstained formalin-fixed paraffin-embedded thin sections
  * All other general (primary or relapsed) cases

    * 10 unstained formalin-fixed paraffin-embedded thin sections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rhabdomyosarcoma enrolled on COG-D9902.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Molecular response | Up to 1 year
Novel pathway/biomarkers detected within clinically annotated patient tumor tissue samples | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pelloski, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States